CLINICAL TRIAL: NCT05391646
Title: Pulmonary Embolism Registry
Acronym: PER
Status: Not yet recruiting | Type: Observational
Sponsor: Universidade do Porto (Other)
Collaborators: Unidade Local de Saúde de Matosinhos, EPE (Other); Centro Hospitalar Universitário do Porto (Unknown); Centro Hospitalar de Vila Nova de Gaia/Espinho, E.P.E. (Other Government); Hospital da Luz, Portugal (Other); Hospital Centre Hospitalar de Trás-os-Montes e Alto Douro (Other); Hospital de Braga (Other); Centro Hospitalar de Entre o Douro e Vouga (Other); Unidade Local de Saúde do Alto Minho (Other)
Responsible Party: Sponsor
Other Study IDs: PER2022
Record Dates: First submitted 2022-05-13; First posted 2022-05-26 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary Embolism, Venous Thromboembolism, Chronic Thromboembolic Disease
MeSH Terms: conditions — Pulmonary Embolism; Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute Pulmonary Embolism (PE) is the most serious clinical presentation of venous thromboembolism (VTE), a leading cause of cardiovascular mortality, exceeded only by stroke and myocardial infarction. Chronic thromboembolic pulmonary hypertension (CTEPH) is the most severe chronic form of CTED and it occurs in 2-4% of patients after acute PE.

In Portugal little is known about PE epidemiology and its outcomes, including complications like CTED. The main goal of this study is, therefore, to understand PE epidemiology and complications in the northern region of Portugal. This information can enable the organization of a structured health care network that can potentially benefit all PE patients.

ELIGIBILITY:
Inclusion Criteria:

* Acute symptomatic or asymptomatic PE,
* Age >18 years,
* Availability of a minimum data set for PE and a minimum of 3-months follow-up for the primary objective and 36-months for the secondary one. Except for patients who died prior to the 3 or 36 months follow-up.

Exclusion Criteria:

* Enrolment of the patient in any treatment trial in a blinded fashion,
* Lack or withdrawal of patient´s consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The PERR is a prospective multicentric observational study of consecutive patients with confirmed PE by computed tomographic pulmonary angiography or ventilation-perfusion lung scan.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-10-31 (Estimated); Primary Completion 2023-12-16 (Estimated); Study Completion 2026-06-16 (Estimated)

PRIMARY OUTCOMES:
Determine Pulmonary Embolism (PE) prevalence in Portugal | From date of inclusion until the end of the study currently planned (3 to 5 years)
  Number cases per year
Identification of Pulmonary Embolism (PE) risk factors and comorbidities | From date of inclusion until the end of the study currently planned (3 to 5 years)
  Frequency of risk factors and comorbidities
Determine Pulmonary Embolism (PE) clinical management. | From date of inclusion until the end of the study currently planned (3 to 5 years)
  Identification of diagnostic of diagnostic and treatment profile

SECONDARY OUTCOMES:
Access incidence rate of Chronic Thromboembolic Disease (CTED) with or without pulmonary hypertension after acute PE. | From 6 months after date of inclusion until the end of the study currently planned (2 to 5 years)
  ratio between the number of patients with CTED with or without pulmonary hypertension and total number of patients with PE

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Guedes, MD, PhDc, Principal Investigator — Universidade do Porto